CLINICAL TRIAL: NCT07241546
Title: A Randomized, Double-blind, Placebo-controlled Phase 2a Study of ARO-RAGE Inhalation Solution to Assess Efficacy on Small Airway Dysfunction in Allergen-induced Mild Asthma
Brief Title: Study of Inhaled ARO-RAGE in Allergen-induced Mild Asthma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARORAGE-2001
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-RAGE (Experimental): ARO-RAGE inhalation
  Interventions: Drug: ARO-RAGE
- Placebo (Placebo Comparator): Normal saline (0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-RAGE — Inhalation of nebulized solution
  Arms: ARO-RAGE
Drug: Placebo — Calculated volume to match active treatment by inhalation of nebulized solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the impact of inhaled ARO-RAGE on the late asthmatic response (LAR) following an inhaled allergen challenge in participants with mild atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, mild atopic asthma (FEV1 ≥70% predicted)
* Established allergy confirmed by positive skin prick test at screening
* Willing and able to perform lung function tests and other study-related procedures
* Participants of childbearing potential must consent to use a method of highly-effective contraception in addition to a condom during the study and for at least 90 days following the end of study or last investigational product administration, whichever is later

Exclusion Criteria:

* Concomitant diagnosis of a clinically important pulmonary disease other than asthma
* Use of corticosteroids, immunosuppressives, or anti-inflammatory medications that interfere with inhaled challenges or inflammation, or chronic use of any other medication for treatment of allergic asthma
* History or current medical condition contraindicating methacholine challenge

Note: Additional inclusion/exclusion criteria may apply per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Over Time in Maximum Area of Reactance | Baseline through Day 58

SECONDARY OUTCOMES:
Change from Baseline Over Time in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve | Baseline through Day 58
Change from Baseline Over Time in Maximum Change in Small Airway Reactance | Baseline through Day 58
Number of Participants with Treatment-Emergent Adverse Events | Up to Day 113, End of Study

IPD SHARING:
Plan to Share IPD: No